CLINICAL TRIAL: NCT03578367
Title: A Phase 2, Multi-center, Open-label, Randomized Study of Oral Asciminib Added to Imatinib Versus Continued Imatinib Versus Switch to Nilotinib in Patients With CML-CP Who Have Been Previously Treated With Imatinib and Have Not Achieved Deep Molecular Response
Brief Title: Study of Efficacy and Safety of Asciminib in Combination With Imatinib in Patients With Chronic Myeloid Leukemia in Chronic Phase (CML-CP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CABL001E2201; 2018-001594-24 (EudraCT Number); 2024-515040-23-00 (Other: EU CTIS)
Record Dates: First submitted 2018-06-15; First posted 2018-07-06 (Actual); Results first posted 2025-02-14 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: CML; Chronic Myelogenous Leukemia; Leukemia, Myeloid Chronic; Hematologic Diseases
Keywords: CML; Chronic Myelogenous Leukemia; leukemia, myeloid chronic; Hematologic Diseases; Asciminib; ABL001; Imatinib; Nilotinib; deep molecular response; DMR; Ph+ CML; chronic phase; cancer of the white blood cells; tyrosine kinase inhibitor; leukemia, myeloid; leukemia; CML with Ph+
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Hematologic Diseases; Leukemia, Myeloid; Leukemia | interventions — asciminib; Imatinib Mesylate; nilotinib

STUDY DESIGN:
Intervention Model Description: Treatment arms 1 - 4 randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Asciminib 60mg QD + Imatinib 400mg QD (Experimental): Asciminib 60 mg taken once daily in combination with Imatinib 400 mg taken once daily
  Interventions: Drug: Asciminib add-on; Drug: Imatinib
- Asciminib 40mg QD + Imatinib 400mg QD (Experimental): Asciminib 40 mg taken once daily in combination with Imatinib 400 mg taken once daily
  Interventions: Drug: Asciminib add-on; Drug: Imatinib
- Imatinib 400mg QD (Active Comparator): Imatinib 400 mg taken once daily
  Interventions: Drug: Imatinib
- Nilotinib 300mg BID (Active Comparator): Nilotinib 300 mg taken twice daily
  Interventions: Drug: Nilotinib

INTERVENTIONS:
Drug: Asciminib add-on — Asciminib 60 mg or 40 mg taken orally once daily.
  Other Names: ABL001 (asciminib)
  Arms: Asciminib 40mg QD + Imatinib 400mg QD; Asciminib 60mg QD + Imatinib 400mg QD
Drug: Imatinib — Imatinib 400 mg taken orally once daily
  Other Names: STI571
  Arms: Asciminib 40mg QD + Imatinib 400mg QD; Asciminib 60mg QD + Imatinib 400mg QD; Imatinib 400mg QD
Drug: Nilotinib — Nilotinib 300 mg taken orally twice daily (total daily dose of 600 mg)
  Other Names: AMN107
  Arms: Nilotinib 300mg BID

SUMMARY:
To evaluate efficacy, safety and pharmacokinetic profile of asciminib 40mg+imatinib or asciminib 60mg+imatinib versus continued imatinib and versus nilotinib versus asciminib 80mg in pre-treated patients with Chronic Myeloid Leukemia in chronic phase (CML-CP)

DETAILED DESCRIPTION:
The study is a Phase 2, multi-center, open-label, randomized study of asciminib in two different doses (40 mg or 60 mg) in combination with imatinib 400 mg versus continued imatinib versus switch to nilotinib in Participants with chronic myeloid leukemia in chronic phase (CML-CP) who have been previously treated with imatinib first line therapy for at least one year and have not achieved deep molecular response (DMR). Eligible participants were randomized 1:1:1:1 to receive asciminib 60 mg once daily (QD) as add-on therapy to imatinib 400 mg QD, or 40 mg QD as add-on therapy to imatinib 400 mg QD, or to continue imatinib 400 mg QD, or to switch to nilotinib 300 mg twice a day (BID).

Participants on the imatinib continuation arm who had not achieved MR4.5 at 48 weeks were allowed to cross-over (CO) to receive the add-on treatment within 4 weeks after week 48 visit to receive the asciminib 60 mg combination add-on treatment, as this dose provided higher exposure. The cross-over is at the discretion of the investigator and the participant. Apart from a polymerase chain reaction (PCR) result of below MR4.5 at Week 48 visit, there are no other entry criteria for the cross-over part. Participants on nilotinib are not allowed to cross- over to receive the add-on treatment.

Participants on the study will continue on the allocated treatment until treatment failure, intolerability, or for up to 96 weeks (in arms 1 to 4) after the last participant received the first dose of treatment. After the last dose received, every participant will be followed up for safety for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 18 years of age with a confirmed diagnosis of Chronic Myeloid Leukemia in chronic phase (CML-CP).
* Minimum of one year (12 calendar months) treatment with imatinib first line for CML-CP (patients have to be on imatinib 300mg or 400 mg QD at randomization

For Korea only:

(i)a minimum of one year (12 calendar months) of prior treatment with imatinib for patients with BCR-ABL levels > 0.1%, ≤ 1% IS at the time of randomization.

(ii) a minimum of two years (24 calendar months) of prior treatment with imatinib for patients with BCR-ABL levels > 0.01%, ≤ 0.1% IS at the time of randomization.

* BCR-ABL1 levels > 0.01% IS (International Scale) and ≤ 1% IS at the time of randomization as confirmed with a central assessment at screening; patients must not have achieved deep molecular response (MR4 IS) confirmed by 2 consecutive tests at any time during prior imatinib treatment. An isolated, single test result with BCR-ABL1 levels < 0.01 % (MR4 IS) is allowed, however, it should not have been observed within the 9 months prior to randomization
* Patient must meet the following laboratory values before randomization:
* Absolute Neutrophil Count ≥ 1.5 x 10E9/L
* Platelets ≥ 75 x 10E9/L
* Hemoglobin ≥ 9 g/dL
* Serum creatinine < 1.5 mg/dL
* Total bilirubin ≤ 1.5 x ULN (Upper Limit of Normal) except for patients with Gilbert's syndrome who may only be included with total bilirubin ≤ 3.0 x ULN
* Aspartate transaminase (AST) ≤ 3.0 x ULN
* Alanine transaminase (ALT) ≤ 3.0 x ULN
* Alkaline phosphatase ≤ 2.5 x ULN
* Serum lipase ≤ 1.5 x ULN
* Participantss must have the following laboratory values ≥ Lower Limit of Normal or corrected to within normal limits with supplements prior to randomization: potassium increase of up to 6.0 mmol/L is acceptable if associated with creatinine clearance within normal limits ; calcium increase of up to 12.5 mg/dl or 3.1 mmol/L is acceptable if associated with creatinine clearance* within normal limits) ; magnesium increase up to 3.0 mg/dL or 1.23 mmol/L if associated with creatinine clearance within normal limits.

Key Exclusion Criteria:

* Treatment failure according to European Leukemia Network (ELN) criteria 2013 during imatinib treatment.
* Known second chronic phase of CML after previous progression to Accelerated Phase (AP)/Blast Crisis (BC).
* Previous treatment with any tyrosine kinese inhibitors (TKIs) other than imatinib.
* History or current diagnosis of ECG abnormalities indicating significant risk or safety for participants participating in the study such as:
* History of myocardial infarction, angina pectoris, coronary artery bypass graft within 6 months prior to randomization
* Concomitant clinically significant arrhythmias
* Resting QTcF ≥ 450 msec (male) or ≥ 460 msec (female) prior to randomization
* Long QT syndrome, family history of idiopathic sudden death or congenital long QT syndrome, or any of the following:

  * Risk factors for Torsades de Pointes
  * Concomitant medications with a "known" risk of Torsades de Pointes
  * inability to determine the QTcF interval 5. Severe and/or uncontrolled concurrent medical disease that in the opinion of the investigator could cause unacceptable safety risks or compromise compliance with the protocol (e.g. uncontrolled diabetes, active or uncontrolled infection, uncontrolled clinically significant hyperlipidemia and high serum amylase) 6. History of acute pancreatitis within 1 year prior to randomization or medical history of chronic pancreatitis; on-going acute liver disease or history of chronic liver disease 7. History of other active malignancy within 3 years prior to randomization with the exception of basal cell skin cancer, indolent prostate cancer and carcinoma in situ treated curatively.

Other protocol defined inclusion/exclusion may apply.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2018-11-22 (Actual); Primary Completion 2021-11-08 (Actual); Study Completion 2025-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (28):
- United States (2):
  - Georgia Regents University, Augusta, Georgia
  - Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
- Novartis Investigative Site, Vienna, Austria
- Novartis Investigative Site, Montreal, Quebec, Canada
- Novartis Investigative Site, Brno, Czechia
- Novartis Investigative Site, Copenhagen, Denmark
- Novartis Investigative Site, Bordeaux, France
- Novartis Investigative Site, Dresden, Germany
- Italy (2):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Roma, RM
- Poland (3):
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Wroclaw
- Portugal (2):
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Porto
- Russia (2):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
- South Korea (2):
  - Novartis Investigative Site, Uijeongbu-si, Gyeonggi-do
  - Novartis Investigative Site, Seoul, Seocho Gu
- Spain (4):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Badalona, Catalonia
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Valencia
- Taiwan (2):
  - Novartis Investigative Site, Changhua
  - Novartis Investigative Site, Taoyuan District
- United Kingdom (3):
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com.
URL: https://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Hughes TP, Saglio G, Geissler J, Kim DW, Lomaia E, Mayer J, Turkina A, Kapoor S, Cardoso AP, Nieman B, Quenet S, Cortes JE. Asciminib add-on to imatinib demonstrates sustained high rates of ongoing therapy and deep molecular responses with prolonged follow-up in the ASC4MORE study. J Hematol Oncol. 2024 Dec 18;17(1):125. doi: 10.1186/s13045-024-01642-6. PMID 39696526

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All the participants were enrolled at 29 sites.
Pre-assignment Details: A total of 84 participants were planned to be randomized to arms 1 to 4.
Period: Overall Study
Arm/Group | Asciminib 40mg QD + Imatinib 400mg QD | Asciminib 60mg QD + Imatinib 400mg QD | Imatinib 400mg QD | Nilotinib 300mg BID
Started | 21 | 21 | 21 | 21
Treated | 21 | 21 | 20 | 21
Discontinued From Treatment | 3 | 5 | 15 | 8
Entered Safety Follow-up | 0 | 2 | 1 | 6
Discontinued Safety Follow-up | 0 | 1 | 1 | 5
Completed (Completed = Patients ongoing on treatment at the time of the primary analysis cut-off) | 18 | 16 | 5 | 13
Not Completed | 3 | 5 | 16 | 8
Not completed — Adverse Event | 0 | 3 | 0 | 5
Not completed — Withdrawal by Subject | 2 | 2 | 1 | 3
Not completed — Physician Decision | 0 | 0 | 14 | 0
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Not treated | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis set (FAs):
Groups:
- Total: Total of all reporting groups
Arm/Group | Asciminib 40mg QD + Imatinib 400mg QD | Asciminib 60mg QD + Imatinib 400mg QD | Imatinib 400mg QD | Nilotinib 300mg BID | Total
Number analyzed (Participants) | 21 | 21 | 21 | 21 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.4 (16.87) | 43.7 (15.72) | 51.0 (15.46) | 44.4 (13.12) | 46.6 (15.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 5 | 6 | 24
  Male | 13 | 16 | 16 | 15 | 60
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 17 | 15 | 19 | 16 | 67
  Chinese | 0 | 0 | 0 | 1 | 1
  Indian | 0 | 1 | 0 | 0 | 1
  Korean | 1 | 2 | 1 | 1 | 5
  Missing Asian | 3 | 1 | 0 | 2 | 6
  Missing - Overall | 0 | 2 | 1 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Molecular Response (MR)^4.5 Rate at 48 Weeks
Description: Percentage of participants still treated with the randomized treatment at 48 weeks and are in MR4.5 (BCR::ABL1 ratio of ≤ 0.0032%) at 48 weeks (± assessment window), among all participants in the asciminib add-on arms vs imatinib arm.
Time Frame: at Week 48
Population: Full analysis set (FAS): The Full Analysis Set comprised all participants to whom study treatment has been assigned by randomization.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Asciminib 40mg QD + Imatinib 400mg QD | Asciminib 60mg QD + Imatinib 400mg QD | Imatinib 400mg QD
Number analyzed (Participants) | 21 | 21 | 21
Percentage of participants | 19.0 [6.8 to 38.4] | 28.6 [13.2 to 48.7] | 0.0 [0.0 to 13.3]
Statistical Analysis 1: Comparison: Asciminib 40mg QD + Imatinib 400mg QD vs Imatinib 400mg QD; Test type: Other — No test performed; Risk Difference (RD) = 19.5, 90% CI 2-sided [5.0 to 33.1]
Statistical Analysis 2: Comparison: Asciminib 60mg QD + Imatinib 400mg QD vs Imatinib 400mg QD; Test type: Other — No test performed; Risk Difference (RD) = 28.57, 90% CI 2-sided [12.4 to 44.8]

2. Secondary Outcome: Rate of MR^4.5 at 48 Weeks
Description: Percentage of participants in MR^4.5 (BCR-ABL1 ratio of ≤ 0.0032%) at 48 weeks in asciminib add-on arms vs nilotinib arm.
Time Frame: at Week 48
Population: FAS: The FAS comprised all participants to whom study treatment has been assigned by randomization.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Asciminib 40mg QD + Imatinib 400mg QD | Asciminib 60mg QD + Imatinib 400mg QD | Nilotinib 300mg BID
Number analyzed (Participants) | 21 | 21 | 21
Percentage of participants | 19.0 [6.8 to 38.4] | 28.6 [13.2 to 48.7] | 4.8 [0.2 to 20.7]
Statistical Analysis 1: Comparison: Asciminib 40mg QD + Imatinib 400mg QD vs Nilotinib 300mg BID; Test type: Other — No test performed; Risk Difference (RD) = 14.29, 90% CI 2-sided [-1.7 to 30.3]
Statistical Analysis 2: Comparison: Asciminib 60mg QD + Imatinib 400mg QD vs Nilotinib 300mg BID; Test type: Other — No test performed; Risk Difference (RD) = 23.81, 90% CI 2-sided [5.9 to 41.7]

3. Secondary Outcome: Rate of MR^4.5 by 48 Weeks
Description: Best observed MR^4.5 rate (BCR-ABL1 ratio of ≤ 0.0032%) up to 48 weeks. This includes the percentage of participants who achieved MR 4.5 anytime up to 48 weeks.
Time Frame: by 48 weeks
Population: FAS: The FAS comprised all participants to whom study treatment has been assigned by randomization.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Asciminib 60mg QD + Imatinib 400mg QD | Asciminib 40mg QD + Imatinib 400mg QD | Imatinib 400mg QD | Nilotinib 300mg BID
Number analyzed (Participants) | 21 | 21 | 21 | 21
Percentage of participants | 19.0 [6.8 to 38.4] | 28.6 [13.2 to 48.7] | 0 [0.0 to 13.3] | 14.3 [4.0 to 32.9]

4. Secondary Outcome: Rate of MR^4.5 at 96 Weeks
Description: Percentage of participants with MR^4.5 rate (BCR-ABL1 ratio of ≤ 0.0032%) at 96 weeks
Time Frame: at 96 weeks
Reporting Status: Not Posted, anticipated posting 2026-02

5. Secondary Outcome: Rate of MR^4.5 by 96 Weeks
Description: Best observed MR4.5 rate (BCR-ABL1 ratio of ≤ 0.0032%) up to 96 weeks
Time Frame: by 96 weeks
Reporting Status: Not Posted, anticipated posting 2026-02

6. Secondary Outcome: Sustained MR^4.5 From 48 Weeks Until 96 Weeks
Description: Percentage of participants who are in MR^4.5 at 48 weeks and 96 weeks and who have no loss of MR^4.5 in between those 2 time points.
Time Frame: at 96 weeks
Reporting Status: Not Posted, anticipated posting 2026-02

7. Secondary Outcome: Time to MR^4.5
Description: Time to MR^4.5 is the time from first dose to first MR^4.5 (BCR-ABL1 ratio of ≤ 0.0032%) computed only for participants who achieved MR^4.5.
Time Frame: 96/48 weeks after the last rand./enrolled (asciminib 80mg cohort) participant received the first study dose
Reporting Status: Not Posted, anticipated posting 2026-02

8. Secondary Outcome: Duration of MR^4.5
Description: Time from first MR^4.5 (BCR-ABL1 ratio of ≤ 0.0032%) until loss of MR^4.5.
Time Frame: 96/48 weeks after the last rand./enrolled (asciminib 80mg cohort) participant received the first study dose
Reporting Status: Not Posted, anticipated posting 2026-02

9. Secondary Outcome: Pharmacokinetic Profile of Asciminib and Imatinib When Administered in Combination - Cmax
Description: The maximum (peak) observed drug concentration after dose administration
Time Frame: up to 96 weeks
Reporting Status: Not Posted, anticipated posting 2026-02

10. Secondary Outcome: Pharmacokinetic Profile of Asciminib and Imatinib When Administered in Combination - Tmax
Description: The time to reach maximum (peak) drug concentration after dose administration
Time Frame: up to 96 weeks
Reporting Status: Not Posted, anticipated posting 2026-02

11. Secondary Outcome: Pharmacokinetic Profile of Asciminib and Imatinib When Administered in Combination - Cmin
Description: Minimum drug concentration
Time Frame: up to 96 weeks
Reporting Status: Not Posted, anticipated posting 2026-02

12. Secondary Outcome: Pharmacokinetic Profile of Asciminib and Imatinib When Administered in Combination - AUClast
Description: The AUC from time zero to the last measurable concentration sampling time (Tlast)
Time Frame: up to 96 weeks
Reporting Status: Not Posted, anticipated posting 2026-02

13. Secondary Outcome: Pharmacokinetic Profile of Asciminib and Imatinib When Administered in Combination - AUCtau
Description: The AUC calculated to the end of a dosing interval (tau) at steady-state
Time Frame: up to 96 weeks
Reporting Status: Not Posted, anticipated posting 2026-02

14. Secondary Outcome: MR^4.5 Rate at 48 Weeks
Description: The percentage of participants on asciminib 80mg QD with MR^4.5 (BCR-ABL1 ratio of ≤ 0.0032%) at 48 weeks
Time Frame: at 48 weeks
Reporting Status: Not Posted, anticipated posting 2026-02

15. Secondary Outcome: Pharmacokinetic Profile of Asciminib 80mg QD - Cmax
Description: The maximum (peak) observed drug concentration after dose administration
Time Frame: up to 48 weeks
Reporting Status: Not Posted, anticipated posting 2026-02

16. Secondary Outcome: Pharmacokinetic Profile of Asciminib 80mg QD - Tmax
Description: The time to reach maximum (peak) drug concentration after dose administration
Time Frame: up to 48 weeks
Reporting Status: Not Posted, anticipated posting 2026-02

17. Secondary Outcome: Pharmacokinetic Profile of Asciminib 80mg QD - Cmin
Description: Minimum drug concentration
Time Frame: up to 48 weeks
Reporting Status: Not Posted, anticipated posting 2026-02

18. Secondary Outcome: Pharmacokinetic Profile of Asciminib 80mg QD - AUClast
Description: The AUC from time zero to the last measurable concentration sampling time (Tlast)
Time Frame: up to 48 weeks
Reporting Status: Not Posted, anticipated posting 2026-02

19. Secondary Outcome: Pharmacokinetic Profile of Asciminib 80mg QD - AUCtau
Description: The AUC calculated to the end of a dosing interval (tau) at steady-state
Time Frame: up to 48 weeks
Reporting Status: Not Posted, anticipated posting 2026-02

ADVERSE EVENTS:
Time Frame: AEs & on-treatment deaths were collected from the first dose of study treatment up to 30 days after last dose of study medication. The maximum duration of treatment exposure was 160 weeks for asciminib 40 mg + imatinib, 148 weeks for asciminib 60 mg + imatinib, 142 weeks for imatinib and 146 weeks for nilotinib.
Description: Any sign or symptom that occurs during the study treatment plus the 30 days post treatment. Adverse events were analyzed in the Safety analysis set, which comprises all patients who received at least one dose of study treatment.
Arm/Group | Asciminib 40mg QD + Imatinib 400mg QD | Asciminib 60mg QD + Imatinib 400mg QD | Imatinib 400mg QD | Nilotinib 300mg BID
All-Cause Mortality (participants affected / at risk) | 1/21 | 0/21 | 0/20 | 0/21
Serious Adverse Events (participants affected / at risk) | 3/21 | 3/21 | 0/20 | 5/21
Other Adverse Events (participants affected / at risk) | 19/21 | 17/21 | 13/20 | 20/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Asciminib 40mg QD + Imatinib 400mg QD (N=21) | Asciminib 60mg QD + Imatinib 400mg QD (N=21) | Imatinib 400mg QD (N=20) | Nilotinib 300mg BID (N=21)
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 0
Appendiceal mucocoele (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Asciminib 40mg QD + Imatinib 400mg QD (N=21) | Asciminib 60mg QD + Imatinib 400mg QD (N=21) | Imatinib 400mg QD (N=20) | Nilotinib 300mg BID (N=21)
Neutropenia (Blood and lymphatic system disorders) | 2 | 1 | 0 | 0
Gilbert's syndrome (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 3
Tinnitus (Ear and labyrinth disorders) | 2 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 5 | 2 | 3 | 1
Nausea (Gastrointestinal disorders) | 7 | 3 | 2 | 3
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 2 | 1 | 2 | 1
Fatigue (General disorders) | 3 | 2 | 0 | 2
COVID-19 (Infections and infestations) | 3 | 2 | 2 | 2
Conjunctivitis (Infections and infestations) | 2 | 0 | 1 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 3
Urinary tract infection (Infections and infestations) | 3 | 1 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 0 | 5
Amylase increased (Investigations) | 1 | 1 | 2 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 3
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 3
Blood cholesterol increased (Investigations) | 0 | 1 | 0 | 3
Blood creatine phosphokinase increased (Investigations) | 1 | 2 | 2 | 1
Blood creatinine increased (Investigations) | 2 | 2 | 0 | 0
Blood phosphorus decreased (Investigations) | 2 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 2
Lipase increased (Investigations) | 3 | 3 | 3 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 2 | 3 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 1 | 1 | 2
Headache (Nervous system disorders) | 3 | 1 | 0 | 2
Paraesthesia (Nervous system disorders) | 0 | 1 | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 3 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 3 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 1 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 8
Hypertension (Vascular disorders) | 1 | 0 | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e., data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2023-08-24): https://cdn.clinicaltrials.gov/large-docs/67/NCT03578367/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-25): https://cdn.clinicaltrials.gov/large-docs/67/NCT03578367/SAP_001.pdf